CLINICAL TRIAL: NCT03521674
Title: Comparison of Foley Catheter and Double-balloon Catheter in Second Trimester Pregnancy Termination
Brief Title: Foley Catheter vs Double-balloon Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Berna Aslan Cetin, Md, ObGYN, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/8
Record Dates: First submitted 2018-04-30; First posted 2018-05-11 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Pregnancy Termination; Catheter
Keywords: second trimester pregnancy termination; double-balloon catheter; foley catheter
MeSH Terms: interventions — Abortion, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Foley catheter (Other): Foley catheter will be inserted through the cervical os and it will be filled with 40 ml saline. After insertion gentle traction will be applied for cervical ripening. Pregnancy termination will be achieved.
  Interventions: Device: pregnancy termination
- Double-balloon catheter (Other): Double-balloon catheter will be inserted through the cervical os and both baloons will be filled with 40 ml saline. No traction will be applied. Pregnancy termination will be achieved.
  Interventions: Device: pregnancy termination

INTERVENTIONS:
Device: pregnancy termination — Second trimester pregnancy termination for fetal anomali or in utero mord fetus will be done

SUMMARY:
The efficiency of double-balloon and Foley catheters in the second trimester medical termination of pregnancies will be compared.

DETAILED DESCRIPTION:
Women will be randomised into two groups. Foley catheter was applied to one group and double balloon catheter to the other group. After catheter expulsion or if the catheters did not spontaneously expulsed after 24 hours, i.v. oxytocin infusion will be started. Abortions will be considered successful if there will be no need of another method for abortion.

ELIGIBILITY:
Inclusion Criteria:

* pregnancy termination, gestational age from 14-24 weeks

Exclusion Criteria:

* multiple gestation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — second trimester pregnancies
Enrollment: 100 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
induction termination interval | during procedure
  time from induction to pregnancy termination

CONTACTS AND LOCATIONS:
Overall Officials: Berna Aslan Çein, Principal Investigator — KSSTRH
Locations (1):
- Kanuni SSTRH, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No